CLINICAL TRIAL: NCT03497052
Title: Blastocyst Developmental Rate in Two Different Single Step Culture Media: a Sibling Oocyte Prospective Non-interventional Study
Brief Title: Culture Media and Blastocyst Development
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinica Valle Giulia (Other)
Responsible Party: Sponsor
Other Study IDs: CVG11112017
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Embryo Development
Keywords: IVF culture media; Blastocyst; Time-lapse microscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Oocytes and embryos will be cultured in GEMS single step medium (in vitro culture in medium 1)
  Interventions: Other: In vitro culture in medium 1
- Group 2: Oocytes and embryos will be cultured in IRVINE single step medium (in vitro culture in medium 2)
  Interventions: Other: In vitro culture in medium 2

INTERVENTIONS:
Other: In vitro culture in medium 1 — Oocytes and embryos will be cultured in GEMS media (single step media) up to blastocyst stage.Standard IVF culture will be performed in a time lapse incubator. No drugs will be used.
  Groups: Group 1
Other: In vitro culture in medium 2 — Oocytes will be cultured in IRVINE media (single step media) up to blastocyst stage.Standard IVF culture will be performed in a time lapse incubator. No drugs will be used.
  Groups: Group 2

SUMMARY:
The aim of this non-interventional study is to compare the blastulation rate per fertilized oocyte in two different single step culture media commercially available (GEMS and Irvine culture media).

DETAILED DESCRIPTION:
SUMMARY:

In ART procedures, blastocyst transfer can be considered the most physiological situation, as the embryo is placed in the uterine cavity at a stage most similar to that which occurs in nature. These potential benefits have induced more and more centres to move from cleavage stage to blastocyst stage embryo transfer all over the world (Maheshwari et al., 2016). Despite this, there are also some potential disadvantages. This approach decreases the total number of usable embryos (defined as those available for transfer or cryopreservation) (Glujovsky et al., 2016). Some concerns regarding the safety of this approach have also been raised. In particular, the extended duration of the in vitro culture may have long-term effect in the embryo development. In a recent meta-analysis, blastocyst stage transfer was in fact associated with increased risks of preterm birth (<37 weeks), very preterm birth (<32 weeks), large for gestational age and perinatal mortality, although the latter was only identified from one study. Conversely, blastocyst transfer was associated with a decrease in the risk of small for gestational age and vanishing twins, although this latter was reported by only one study (Martins et al., 2017).

Culture media plays a crucial role in this context. Two distinct approaches aimed at supporting embryo development to the blastocyst stage have been proposed: the "back to nature" sequential approach and the "let the embryo choose" single medium approach (Summers et al., 2003; Machtinger et al., 2012, Quinn 2012).

Sequential culture media system is designed to meet identified changing metabolic and nutritional requirements of the developing embryo from day 1 to day 5 (Gardner et al. 1996, 1997, 1998, 1999). With this approach, embryos are grown up to day 3 in a first medium and then, at the cleavage stage, are moved to a second one. The goal is to expose the embryos to stage-specific media, designed to reflect observed changes in concentrations of pyruvate, lactate, and glucose in the Fallopian tube versus the uterus (Gardner et al., 1996).

On the other hand, single culture media aim at allowing developing embryos to choose the nutrients they require, while at the same time minimizing stress from exposure to an abrupt change in their culture environment on day 3. Single media can be used with a medium change on day 3, or in a single-step uninterrupted culture, in which there is no medium refreshing on day 3 [Biggers et al., 2008]. Available data comparing the performance of single vs. sequential culture media suggest that both types of media seem to provide similar support to the developing embryo (Sfontouris et al., 2017).

Aim of the study and design

The aim of this non-interventional study is to compare the blastulation rate per fertilized oocyte in two different single step culture media commercially available (GEMS and Irvine culture media).

Oocyte collection

Consecutive egg collection will be performed (with inclusion of oocytes coming from woman not older than 42 years of age, presenting between 4 and 8 normal appearing MII oocytes and undergoing ICSI treatment with ejaculated sperm in the Centre for Reproductive Medicine GENERA in Rome). To exclude potential negative paternal effect on blastulation rate, all oocytes coming from couples with surgically extracted spermatozoa and very severe oligoastenoteratozoospermia (motile sperm count <500.000/ml after preparation) will be excluded. Oocytes coming from patients enrolled in PGD program for monogenic diseases or structural chromosomal abnormalities will be excluded too.

It is estimated, based centre experience, the study will last for 18 months. The informed consent is the GENERA standard format in ordinary use. The study will be approved by the Institutional Review Board of the Clinic.

Oocyte denudation, evaluation and injection All the procedures will be performed according to standard practice without any kind of intervention.

Just after the pick-up procedure, oocytes will be denuded from the cumulus oophorus by a brief exposure to 40 IU/ml hyaluronidase solution followed by mechanical removal of the corona radiata with the use of plastic pipettes of defined diameters in a controlled temperature environment. This procedure will be performed between 37 and 40 hours post hCG administration. Metaphase II (MII) oocytes will be then separated from the immature oocytes and evaluated at the stereomicroscope. Those with severe morphological abnormalities will be considered of lower quality (according to Rienzi et al., 2008) and will thus be excluded from comparison. All the MII oocyte will be placed in the same Petri Dish.

Using randomization tables, oocytes from each patient will be randomly split in two groups that will be independently inseminated and subsequently kept in 2 single step culture media, GEMS (GERI Medium) and Irvine (Continuous Single Culture Complete with HSA). Oocytes will be subjected to ICSI using previously described techniques and instrumentations (Rienzi et al., 1998). To be able to follow the developmental progression of individual oocyte, inseminated oocytes from each group will be cultured in separate dishes and each individual oocyte will be identified according to its position within the dish microwells. Embryo culture will last up to day 5 and will be performed in a time-lapse incubator (GERI, Genea) in hypoxic atmosphere containing 6%CO2 and 5%O2.

Embryo assessment

As per GENERA procedure, detailed analysis of various events during embryo development (syngamy, cleavages, compaction and blastulation) will be assessed using morphokinetic analysis. Various parameters will be assessed: time between the end of the ICSI procedure and syngamy, completion of cleavage to 2, 3, 4, 5 and 8 cells (T2, T3, T4, T5, T8, respectively); length of the first, second and third cell cycle (CC1, CC2, and CC3 respectively) and synchrony in the division from three to four and five to eight cells (S2 and S3, respectively). Standard blastocyst morphological assessment will be performed according to the criteria reported by Gardner and Schoolcraft (1999). In brief, the blastocysts will be evaluated according to the degree of expansion, quality of the inner cell mass (ICM) and of the trophectoderm cells (TE). The ICM is evaluated according to the number of cells, and the degree of compaction, while the TE is evaluated according to the number, dimension of the cells and the appearance of the epithelium (cohesive or loose). Morphokinetic parameters related to blastocyst formation will also be recorded and in particular: initiation of compaction, initiation of blastulation, and completion of blastulation (TSC, TSB, TB, respectively).

Statistical Considerations The primary study endpoint is the blastulation rate, computed as the percentage of fertilized eggs, cultured in either medium, that develop to the blastocyst stage in each half of the cohort. Since only women with between 4 and 8 retrieved oocytes will be eligible, and oocytes from each woman will be randomly split in 2 groups, assuming a fertilization rate of 80% the study population to be analysed will be composed by X*2 (where X is the number of enrolled women) groups of 2+ oocytes, half cultured in one medium and the other cultured in the second medium. The most obvious approach to the analysis of the resulting data is to consider it as a set of X (= number of women) 2x2 tables, where the quantity to be estimated is the odds ratio of blastulation of one medium relative to the other, to be analysed by means of the Mantel Haenszel procedure, with woman as the stratification factor (primary analysis). Assuming an overall blastulation rate of 34% a minimal relevant difference of 7% corresponds to an odds ratio of blastulation of 1.4. In order to detect with alfa=5% (2-sided) and power = 80% an odds ratio of 1.4, approximately 1200 (1182) oocytes need to be included (Hulley et al., 2013) split in 2 groups of equal sizes, that correspond approximately to 160 - 200 women (aprox. 6 oocytes/woman retrieved and considering a fertilization rate 80%).

In secondary exploratory analysis, a logistic model will be fitted to the data with blastulation as the dependent binary variable and woman as stratum, to assess the predictive value of various prognostic factors and the possible interactions between each of them and the culture medium.

ELIGIBILITY:
Inclusion Criteria:

-Woman not older than 42 years of age, presenting between 4 and 8 normal appearing MII oocytes and undergoing ICSI treatment with ejaculated sperm

Exclusion Criteria:

* Men with surgically extracted spermatozoa and very severe oligoastenoteratozoospermia (motile sperm count <500.000/ml after preparation)
* Oocytes coming from patients enrolled in PGT-M (preimplantation genetic testing for monogenic diseases) and PGT-SR (preimplantation genetic testing for structural chromosomal abnormalities) programs.

Max Age: 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Assuming an overall blastulation rate of 34% a minimal relevant difference of 7% corresponds to an odds ratio of blastulation of 1.4. In order to detect with alfa=5% (2-sided) and power = 80% an odds ratio of 1.4, approximately 1200 (1182) oocytes need to be included (Hulley et al., 2013) split in 2 groups of equal sizes, that correspond approximately to 160 - 200 women (aprox. 6 oocytes/woman retrieved and considering a fertilization rate 80%).
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Blastulation rate | 7 days
  The number of embryos reaching the blastocyst stage (day-5, day-6 or day-7 of preimplantation development) per fertilized oocyte (2PN)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Rienzi, MSc, Principal Investigator — Clinica Valle Giulia, G.en.e.r.a. centers for reproductive medicine
Locations (1):
- Clinica Valle Giulia, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Biggers JD, Summers MC. Choosing a culture medium: making informed choices. Fertil Steril. 2008 Sep;90(3):473-83. doi: 10.1016/j.fertnstert.2008.08.010. PMID 18847602
- [Background] Gardner DK, Lane M. Culture and selection of viable blastocysts: a feasible proposition for human IVF? Hum Reprod Update. 1997 Jul-Aug;3(4):367-82. doi: 10.1093/humupd/3.4.367. PMID 9459282
- [Background] 3. Gardner D, Schoolcraft W. In vitro culture of the human blastocyst. In: Jansen R, Mortimer D, editors. Towards reproductive certainty: infertility and genetics beyond 1999. Carnforth, UK: Parthenon Publishing; 1999. p. 378-88
- [Background] Gardner DK, Lane M, Calderon I, Leeton J. Environment of the preimplantation human embryo in vivo: metabolite analysis of oviduct and uterine fluids and metabolism of cumulus cells. Fertil Steril. 1996 Feb;65(2):349-53. doi: 10.1016/s0015-0282(16)58097-2. PMID 8566260
- [Background] Gardner DK, Lane M. Culture of viable human blastocysts in defined sequential serum-free media. Hum Reprod. 1998 Jun;13 Suppl 3:148-59; discussion 160. doi: 10.1093/humrep/13.suppl_3.148. PMID 9755421
- [Background] Glujovsky D, Farquhar C, Quinteiro Retamar AM, Alvarez Sedo CR, Blake D. Cleavage stage versus blastocyst stage embryo transfer in assisted reproductive technology. Cochrane Database Syst Rev. 2016 Jun 30;(6):CD002118. doi: 10.1002/14651858.CD002118.pub5. PMID 27357126
- [Background] Machtinger R, Racowsky C. Culture systems: single step. Methods Mol Biol. 2012;912:199-209. doi: 10.1007/978-1-61779-971-6_12. PMID 22829376
- [Background] Martins WP, Nastri CO, Rienzi L, van der Poel SZ, Gracia CR, Racowsky C. Obstetrical and perinatal outcomes following blastocyst transfer compared to cleavage transfer: a systematic review and meta-analysis. Hum Reprod. 2016 Nov;31(11):2561-2569. doi: 10.1093/humrep/dew244. Epub 2016 Oct 7. PMID 27907898
- [Background] Martins WP, Nastri CO, Rienzi L, van der Poel SZ, Gracia C, Racowsky C. Blastocyst vs cleavage-stage embryo transfer: systematic review and meta-analysis of reproductive outcomes. Ultrasound Obstet Gynecol. 2017 May;49(5):583-591. doi: 10.1002/uog.17327. Epub 2017 Apr 10. PMID 27731533
- [Background] Rienzi L, Ubaldi FM, Iacobelli M, Minasi MG, Romano S, Ferrero S, Sapienza F, Baroni E, Litwicka K, Greco E. Significance of metaphase II human oocyte morphology on ICSI outcome. Fertil Steril. 2008 Nov;90(5):1692-700. doi: 10.1016/j.fertnstert.2007.09.024. Epub 2008 Feb 4. PMID 18249393
- [Background] Ubaldi FM, Capalbo A, Colamaria S, Ferrero S, Maggiulli R, Vajta G, Sapienza F, Cimadomo D, Giuliani M, Gravotta E, Vaiarelli A, Rienzi L. Reduction of multiple pregnancies in the advanced maternal age population after implementation of an elective single embryo transfer policy coupled with enhanced embryo selection: pre- and post-intervention study. Hum Reprod. 2015 Sep;30(9):2097-106. doi: 10.1093/humrep/dev159. Epub 2015 Jul 5. PMID 26150408
- [Background] Quinn P. Culture systems: sequential. Methods Mol Biol. 2012;912:211-30. doi: 10.1007/978-1-61779-971-6_13. PMID 22829377
- [Background] Sfontouris IA, Martins WP, Nastri CO, Viana IG, Navarro PA, Raine-Fenning N, van der Poel S, Rienzi L, Racowsky C. Blastocyst culture using single versus sequential media in clinical IVF: a systematic review and meta-analysis of randomized controlled trials. J Assist Reprod Genet. 2016 Oct;33(10):1261-1272. doi: 10.1007/s10815-016-0774-5. Epub 2016 Aug 5. PMID 27491772
- [Background] Summers MC, Biggers JD. Chemically defined media and the culture of mammalian preimplantation embryos: historical perspective and current issues. Hum Reprod Update. 2003 Nov-Dec;9(6):557-82. doi: 10.1093/humupd/dmg039. PMID 14714592
- [Background] 15. Hulley SB, Cummings SR, Browner WS, Grady D, Newman TB. Designing clinical research: an epidemiologic approach. 4th ed. Philadelphia, PA: Lippincott Williams & Wilkins; 2013. Appendix 6B, page 75